CLINICAL TRIAL: NCT04251754
Title: The Acute Promyelocytic Leukaemia Asian Consortium (APL-AC) Project
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: APLAC001
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Acute Promyelocytic Leukemia
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is currently lack of collaborative data on the epidemiology, clinicopathologic features and treatment outcome of newly diagnosed and relapsed APL in Asia. In addition, there is lack of data comparing oral- As2O3-based regimens with other treatment approaches, including intravenous As2O3,in the frontline or relapsed setting. With the long-term data of oral-As2O3 based regimen for APL available from Hong Kong, retrospective and prospective comparison with other treatment approaches in other Asian countries will generate important information to pave the way for widespread application of oral-As2O3 outside Hong Kong.

DETAILED DESCRIPTION:
Acute promyelocytic leukemia (APL) is characterized by t(15;17)(q24;21) and the fusion gene PML-RARA.1 In newly-diagnosed patients, optimal supportive care together with the use of all-trans retinoic acid (ATRA) and chemotherapy results in first complete remission (CR1) in excess of 90% with durable remissions in about 80% of patients.Arsenic trioxide (As2O3) given intravenously (i.v.-As2O3) is highly efficacious for APL in first relapse (R1), inducing second complete remission (CR2) in more than 90% of patients. We have formulated an oral preparation of As2O3 (oral-As2O3), and shown that it is efficacious for APL in R1, giving CR2 rates of more than 90% in both adults and children. For patients in CR2, a 2-year maintenance with oral-As2O3 results in durable remission and long-term survivals in more than 60% and 70% of patients respectively strongly suggesting that hematopoietic stem cell transplantation (HSCT) could be obviated in such patients. With these results, we implemented oral-As2O3 maintenance in CR1 in Hong Kong and demonstrated very favourable overall-survival (OS) and leukemia-free-survival (LFS). This implied that that prolonged oral-As2O3 treatment may prevent relapses.

Meanwhile, i.v.-As2O3 has also been tested in the frontline treatment of newly-diagnosed APL.These studies employed different strategies, recruiting a mixture of low-, intermediate- to high-risk patients and placing i.v.-As2O3 in induction and/or consolidation. During induction, i.v.-As2O3 was combined with ATRA, with additional gemtuzumab ozogamicin (an anti-CD33 immunoconjugate) or chemotherapy. During consolidation, i.v.-As2O3 was combined with conventional chemotherapy. Their results all indicated that frontline use of i.v.-As2O3 in induction and/or consolidation improved the outcome of newly-diagnosed APL patients. However, with quite diverse protocols and the enrollment in some studies of only patients with low to intermediate risks, and in other studies of patients with all risk categories; the optimal strategy of employing i.v.-As2O3 in newly-diagnosed APL remains to be defined. We have tested oral- As2O3 in combination with ATRA, ascorbic acid (AAA) with daunorubicin in both low-risk and high-risk APL with 3 year LFS and OS of both 100%.

With the impressive results of oral-As2O3-based regimen in newly diagnosed and relapsed APL, an important future perspective is the application of this relatively economical and convenient approach to the treatment of patients with APL in Asia and other developing countries around the world where the cost and availability of intravenous formulation of As2O3 is a concern. There is currently lack of collaborative data on the epidemiology, clinicopathologic features and treatment outcome of newly diagnosed and relapsed APL in Asia. In addition, there is lack of data comparing oral- As2O3-based regimens with other treatment approaches, including intravenous As2O3,in the frontline or relapsed setting. With the long-term data of oral-As2O3 based regimen for APL available from Hong Kong, retrospective and prospective comparison with other treatment approaches in other Asian countries will generate important information to pave the way for widespread application of oral-As2O3 outside Hong Kong.

ELIGIBILITY:
Inclusion criteria:

* Patients aged 18 or above
* Acute promyelocytic leukaemia with PML/RARA
* Acute myeloid leukaemia with variant RARA translocation

Exclusion criteria:

-Acute myeloid leukaemia without PML/RARA or variant RARA translocation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a retrospective-prospective cohort study for all patients diagnosed with acute promyelocytic leukaemia since 2010 in Hong Kong and participating countries in Asia.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-02-02 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Survivals | 60 months
  The primary outcome measures in this study include the overall survival (OS) and the relapse-free survival (RFS). OS is defined as the time (in months) from diagnosis to death from any cause (event) or latest follow-up. RFS is defined as the time from first complete remission (CR)/complete remission with incomplete haematological recovery (CRi) to first hamatologic relapse or molecular relapse (R1) (event), death from any cause (event) or latest follow-up (censor). CR, CRi, treatment failure, haematologic relapse are defined according to the 2017 European LeukemiaNet (ELN) recommendations. A molecular relapse is defined as recurrence of measurable residual disease (MRD) by reverse-transcriptase polymerase chain reaction (RT-PCR) or real-time quantitative PCR (qRT PCR). A single MRD positivity must be confirmed by performing the molecular assay within 2 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Harinder Gill, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Medicine, the University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tallman MS, Altman JK. How I treat acute promyelocytic leukemia. Blood. 2009 Dec 10;114(25):5126-35. doi: 10.1182/blood-2009-07-216457. PMID 19797519
- [Result] Tallman MS, Andersen JW, Schiffer CA, Appelbaum FR, Feusner JH, Woods WG, Ogden A, Weinstein H, Shepherd L, Willman C, Bloomfield CD, Rowe JM, Wiernik PH. All-trans retinoic acid in acute promyelocytic leukemia: long-term outcome and prognostic factor analysis from the North American Intergroup protocol. Blood. 2002 Dec 15;100(13):4298-302. doi: 10.1182/blood-2002-02-0632. Epub 2002 Aug 15. PMID 12393590
- [Result] Lengfelder E, Haferlach C, Saussele S, Haferlach T, Schultheis B, Schnittger S, Ludwig WD, Staib P, Aul C, Gruneisen A, Kern W, Reichle A, Serve H, Berdel WE, Braess J, Spiekermann K, Wormann B, Sauerland MC, Heinecke A, Hiddemann W, Hehlmann R, Buchner T; German AML Cooperative Group. High dose ara-C in the treatment of newly diagnosed acute promyelocytic leukemia: long-term results of the German AMLCG. Leukemia. 2009 Dec;23(12):2248-58. doi: 10.1038/leu.2009.183. Epub 2009 Sep 10. PMID 19741727
- [Result] Lo-Coco F, Avvisati G, Vignetti M, Breccia M, Gallo E, Rambaldi A, Paoloni F, Fioritoni G, Ferrara F, Specchia G, Cimino G, Diverio D, Borlenghi E, Martinelli G, Di Raimondo F, Di Bona E, Fazi P, Peta A, Bosi A, Carella AM, Fabbiano F, Pogliani EM, Petti MC, Amadori S, Mandelli F; Italian GIMEMA Cooperative Group. Front-line treatment of acute promyelocytic leukemia with AIDA induction followed by risk-adapted consolidation for adults younger than 61 years: results of the AIDA-2000 trial of the GIMEMA Group. Blood. 2010 Oct 28;116(17):3171-9. doi: 10.1182/blood-2010-03-276196. Epub 2010 Jul 19. PMID 20644121
- [Result] Kelaidi C, Chevret S, De Botton S, Raffoux E, Guerci A, Thomas X, Pigneux A, Lamy T, Rigal-Huguet F, Meyer-Monard S, Chevallier P, Maloisel F, Deconinck E, Ferrant A, Fegueux N, Ifrah N, Sanz M, Dombret H, Fenaux P, Ades L. Improved outcome of acute promyelocytic leukemia with high WBC counts over the last 15 years: the European APL Group experience. J Clin Oncol. 2009 Jun 1;27(16):2668-76. doi: 10.1200/JCO.2008.18.4119. Epub 2009 May 4. PMID 19414681
- [Result] Niu C, Yan H, Yu T, Sun HP, Liu JX, Li XS, Wu W, Zhang FQ, Chen Y, Zhou L, Li JM, Zeng XY, Yang RR, Yuan MM, Ren MY, Gu FY, Cao Q, Gu BW, Su XY, Chen GQ, Xiong SM, Zhang TD, Waxman S, Wang ZY, Chen Z, Hu J, Shen ZX, Chen SJ. Studies on treatment of acute promyelocytic leukemia with arsenic trioxide: remission induction, follow-up, and molecular monitoring in 11 newly diagnosed and 47 relapsed acute promyelocytic leukemia patients. Blood. 1999 Nov 15;94(10):3315-24. PMID 10552940
- [Result] Soignet SL, Frankel SR, Douer D, Tallman MS, Kantarjian H, Calleja E, Stone RM, Kalaycio M, Scheinberg DA, Steinherz P, Sievers EL, Coutre S, Dahlberg S, Ellison R, Warrell RP Jr. United States multicenter study of arsenic trioxide in relapsed acute promyelocytic leukemia. J Clin Oncol. 2001 Sep 15;19(18):3852-60. doi: 10.1200/JCO.2001.19.18.3852. PMID 11559723
- [Result] Au WY, Li CK, Lee V, Yuen HL, Yau J, Chan GC, Ha SY, Kwong YL. Oral arsenic trioxide for relapsed acute promyelocytic leukemia in pediatric patients. Pediatr Blood Cancer. 2012 Apr;58(4):630-2. doi: 10.1002/pbc.23306. Epub 2011 Sep 2. PMID 21898784
- [Result] Gill H, Yim R, Lee HKK, Mak V, Lin SY, Kho B, Yip SF, Lau JSM, Li W, Ip HW, Hwang YY, Chan TSY, Tse E, Au WY, Kumana CR, Kwong YL. Long-term outcome of relapsed acute promyelocytic leukemia treated with oral arsenic trioxide-based reinduction and maintenance regimens: A 15-year prospective study. Cancer. 2018 Jun 1;124(11):2316-2326. doi: 10.1002/cncr.31327. Epub 2018 Mar 26. PMID 29579321
- [Result] Au WY, Kumana CR, Lee HK, Lin SY, Liu H, Yeung DY, Lau JS, Kwong YL. Oral arsenic trioxide-based maintenance regimens for first complete remission of acute promyelocytic leukemia: a 10-year follow-up study. Blood. 2011 Dec 15;118(25):6535-43. doi: 10.1182/blood-2011-05-354530. Epub 2011 Oct 12. PMID 21998212
- [Result] Hu J, Liu YF, Wu CF, Xu F, Shen ZX, Zhu YM, Li JM, Tang W, Zhao WL, Wu W, Sun HP, Chen QS, Chen B, Zhou GB, Zelent A, Waxman S, Wang ZY, Chen SJ, Chen Z. Long-term efficacy and safety of all-trans retinoic acid/arsenic trioxide-based therapy in newly diagnosed acute promyelocytic leukemia. Proc Natl Acad Sci U S A. 2009 Mar 3;106(9):3342-7. doi: 10.1073/pnas.0813280106. Epub 2009 Feb 18. PMID 19225113
- [Result] Lo-Coco F, Avvisati G, Vignetti M, Thiede C, Orlando SM, Iacobelli S, Ferrara F, Fazi P, Cicconi L, Di Bona E, Specchia G, Sica S, Divona M, Levis A, Fiedler W, Cerqui E, Breccia M, Fioritoni G, Salih HR, Cazzola M, Melillo L, Carella AM, Brandts CH, Morra E, von Lilienfeld-Toal M, Hertenstein B, Wattad M, Lubbert M, Hanel M, Schmitz N, Link H, Kropp MG, Rambaldi A, La Nasa G, Luppi M, Ciceri F, Finizio O, Venditti A, Fabbiano F, Dohner K, Sauer M, Ganser A, Amadori S, Mandelli F, Dohner H, Ehninger G, Schlenk RF, Platzbecker U; Gruppo Italiano Malattie Ematologiche dell'Adulto; German-Austrian Acute Myeloid Leukemia Study Group; Study Alliance Leukemia. Retinoic acid and arsenic trioxide for acute promyelocytic leukemia. N Engl J Med. 2013 Jul 11;369(2):111-21. doi: 10.1056/NEJMoa1300874. PMID 23841729
- [Result] Abaza Y, Kantarjian H, Garcia-Manero G, Estey E, Borthakur G, Jabbour E, Faderl S, O'Brien S, Wierda W, Pierce S, Brandt M, McCue D, Luthra R, Patel K, Kornblau S, Kadia T, Daver N, DiNardo C, Jain N, Verstovsek S, Ferrajoli A, Andreeff M, Konopleva M, Estrov Z, Foudray M, McCue D, Cortes J, Ravandi F. Long-term outcome of acute promyelocytic leukemia treated with all-trans-retinoic acid, arsenic trioxide, and gemtuzumab. Blood. 2017 Mar 9;129(10):1275-1283. doi: 10.1182/blood-2016-09-736686. Epub 2016 Dec 21. PMID 28003274
- [Result] Iland HJ, Bradstock K, Supple SG, Catalano A, Collins M, Hertzberg M, Browett P, Grigg A, Firkin F, Hugman A, Reynolds J, Di Iulio J, Tiley C, Taylor K, Filshie R, Seldon M, Taper J, Szer J, Moore J, Bashford J, Seymour JF; Australasian Leukaemia and Lymphoma Group. All-trans-retinoic acid, idarubicin, and IV arsenic trioxide as initial therapy in acute promyelocytic leukemia (APML4). Blood. 2012 Aug 23;120(8):1570-80; quiz 1752. doi: 10.1182/blood-2012-02-410746. Epub 2012 Jun 19. PMID 22715121
- [Result] Platzbecker U, Avvisati G, Cicconi L, Thiede C, Paoloni F, Vignetti M, Ferrara F, Divona M, Albano F, Efficace F, Fazi P, Sborgia M, Di Bona E, Breccia M, Borlenghi E, Cairoli R, Rambaldi A, Melillo L, La Nasa G, Fiedler W, Brossart P, Hertenstein B, Salih HR, Wattad M, Lubbert M, Brandts CH, Hanel M, Rollig C, Schmitz N, Link H, Frairia C, Pogliani EM, Fozza C, D'Arco AM, Di Renzo N, Cortelezzi A, Fabbiano F, Dohner K, Ganser A, Dohner H, Amadori S, Mandelli F, Ehninger G, Schlenk RF, Lo-Coco F. Improved Outcomes With Retinoic Acid and Arsenic Trioxide Compared With Retinoic Acid and Chemotherapy in Non-High-Risk Acute Promyelocytic Leukemia: Final Results of the Randomized Italian-German APL0406 Trial. J Clin Oncol. 2017 Feb 20;35(6):605-612. doi: 10.1200/JCO.2016.67.1982. Epub 2016 Oct 31. PMID 27400939
- [Result] Powell BL, Moser B, Stock W, Gallagher RE, Willman CL, Stone RM, Rowe JM, Coutre S, Feusner JH, Gregory J, Couban S, Appelbaum FR, Tallman MS, Larson RA. Arsenic trioxide improves event-free and overall survival for adults with acute promyelocytic leukemia: North American Leukemia Intergroup Study C9710. Blood. 2010 Nov 11;116(19):3751-7. doi: 10.1182/blood-2010-02-269621. Epub 2010 Aug 12. PMID 20705755
- [Result] Gill H, Kumana CR, Yim R, Hwang YY, Chan TSY, Yip SF, Lee HKK, Mak V, Lau JSM, Chan CC, Kho B, Wong RSM, Li W, Lin SY, Lau CK, Ip HW, Leung RYY, Lam CCK, Kwong YL. Oral arsenic trioxide incorporation into frontline treatment with all-trans retinoic acid and chemotherapy in newly diagnosed acute promyelocytic leukemia: A 5-year prospective study. Cancer. 2019 Sep 1;125(17):3001-3012. doi: 10.1002/cncr.32180. Epub 2019 May 15. PMID 31090936
- [Derived] Gill H, Raghupathy R, Hou HA, Cheng-Hong Tsai X, Tantiworawit A, Ooi MG, Gan GG, Wong CL, Yim R, Chin L, Lee P, Li VWK, Au L, Zhang Q, Leung GMK, Wu TKY, Lee CYY, Chng WJ, Tien HF, Kumana CR, Kwong YL. Acute Promyelocytic Leukemia Asian Consortium study of arsenic trioxide in newly diagnosed patients: impact and outcome. Blood Adv. 2025 Feb 25;9(4):862-876. doi: 10.1182/bloodadvances.2024014999. PMID 39693517
- [Derived] Gill H, Raghupathy R, Lee CYY, Yung Y, Chu HT, Ni MY, Xiao X, Flores FP, Yim R, Lee P, Chin L, Li VWK, Au L, Au WY, Ma ESK, Mohan D, Kumana CR, Kwong YL. Acute promyelocytic leukaemia: population-based study of epidemiology and outcome with ATRA and oral-ATO from 1991 to 2021. BMC Cancer. 2023 Feb 10;23(1):141. doi: 10.1186/s12885-023-10612-z. PMID 36765318